CLINICAL TRIAL: NCT00146432
Title: Prospective, Controlled Pilot Trial: Treatment of Patients in Severe Sepsis and Septic Shock With Immunoadsorption of LPS, IL-6, C5a
Brief Title: Immunoadsorption of LPS, C5a and IL-6 in Severe Sepsis and Septic Shock (ISASS-1)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Research Foundation (Other); adexter GmbH (Industry)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ISASS-1
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Septicemia
MeSH Terms: conditions — Sepsis | interventions — Interleukin-6; Receptor, Anaphylatoxin C5a

INTERVENTIONS:
Procedure: Immunoadsorption of LPS, IL-6 and C5a

SUMMARY:
The purpose of this study is to determine whether immunoadsorption of LPS, Il-6 and C5a reduces systemic hyperinflammation, improves immune function and improves organ function in patients with severe sepsis and septic shock

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe sepsis or septic shock (ACCP/SCCM)
* Presence of 4 SIRS criteria/indicators
* Suspected or proven infection (refer also to: 1.)
* Age 18-80
* APACHE II score > 18
* At least one acute organ dysfunction (renal/pulmonary/hemodynamics/cerebral)

Exclusion Criteria:

* Suspected or proven pregnancy
* Absolute contraindication for anticoagulation (active bleeding)
* Absolute IgA-deficiency
* History of anaphylactic reaction to egg-albumin
* Participants in other clinical trials (<12 wks. prior to study inclusion)

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Petra Reinke, MD, PhD, Principal Investigator — Charite, University Medicine Berlin, Germany
Locations (1):
- Charite University Medicine Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Schefold JC, von Haehling S, Corsepius M, Pohle C, Kruschke P, Zuckermann H, Volk HD, Reinke P. A novel selective extracorporeal intervention in sepsis: immunoadsorption of endotoxin, interleukin 6, and complement-activating product 5a. Shock. 2007 Oct;28(4):418-25. doi: 10.1097/shk.0b013e31804f5921. PMID 17558345
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/18448264?ordinalpos=14&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_DefaultReportPanel.Pubmed_RVDocSum